CLINICAL TRIAL: NCT00816270
Title: Comparison Between Liquid Bandage(2-Octyl-Cyanoacrylate)and Traditional Suture Closure in Upper Lid Blepharoplasty
Brief Title: Liquid Bandage (2-Octyl-Cyanoacrylate) in Upper Lid Blepharoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Experimental results were unsatisfatory compared with control.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Angelino Julio Cariello, Federal University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 1716/07
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Blepharoptosis
Keywords: Blepharoptosis; Dermatochalasis; octyl 2-cyanoacrylate; Suture Techniques; Tissue Adhesive
MeSH Terms: conditions — Blepharoptosis; Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Experimental operatory wound closure with liquid bandage (Johnson & Johnson, Skillman, NJ, USA).
  Interventions: Procedure: Bilateral Upper eyelid blepharoplasty

INTERVENTIONS:
Procedure: Bilateral Upper eyelid blepharoplasty — Bilateral upper lid blepharoplasty was performed on each patient by the same experimented surgeon using a standard technique. One side (right or left upper eyelid) was randomly chosen for experimental closure with liquid bandage and the opposite eyelid served as the control being used a 6/0 nylon continuous sutures.
  Other Names: Liquid bandage (Johnson & Johnson, Skillman, NJ, USA); nylon continuous sutures (Ethicon, Norderstedt, Germany)

SUMMARY:
The aim of this randomized and masked prospective trial is to compare the effectiveness of Liquid Bandage (Octyl-2-Cyanoacrylate) and 6/0 nylon suture as a wound closure device in upper lid blepharoplasty surgery.

DETAILED DESCRIPTION:
Tissue adhesives have been safely used in a variety of surgical procedures for several years. Butyl-2-cyanoacrylate (Histoacryl) and Octyl-2-cyanoacrylate (Dermabond) was also studied for cosmetic blepharoplasty with satisfactory results. Liquid Bandage (Johnson & Johnson, Skillman, NJ, USA) is a more flexible formulation of octyl-2-cyanoacrylate available in many american drugstores for home use. Animal models shown that this product could accelerate the healing of lamellar wounds and studies in humans have demonstrated its safety and effectiveness as an occlusive protective film over cuts, abrasion and wound surgery. Liquid Bandage was also used as a temporary wound barrier in clear corneal cataract surgery with satisfactory applicability. There is no study in the literature using this device in blepharoplasty yet.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 25 years with diagnosis of dermatochalasis who presented surgical indication of primary blepharoplasty.

Exclusion Criteria:

* Prior eyelid surgery
* Concomitant ocular or systemic disease or current use of medications that could interfere in coagulation or wound healing (eg, diabetes mellitus, oral acetyl salicylic acid or corticosteroids)
* Pregnant female
* Known allergy to cyanoacrylate
* Inability to return for follow-up consultations

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The overall cosmetic outcome of wound closure technique (experimental: tissue adhesive Octyl-2-cyanoacrylate versus control: traditional nylon suture). | thirty days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Angelino J Cariello, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Department of Ophthalmology of Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Veloudios A, Kratky V. Cyanoacrylate Tissue Adhesive in Blepharoplasty. Ophthalm Plastic Reconstr Surg 1996;12(2):89-97. Greene D, Koch RJ, Goode RL. Efficacy of Octyl-2-Cyanoacrylate Tissue Glue in Blepharoplasty. Arch Facial Plast Surg 1999;1:292-6. Davis SC, Eaglstein WH, Cazzaniga AL, Mertz PM. An octyl-2-cyanoacrylate formulation speeds healing of partial-thickness wounds. Dermatol Surg 2001;27:783-8.